CLINICAL TRIAL: NCT01932580
Title: Pilot Study of Perioperative Docetaxel, Oxaliplatin, and 5-Fluorouracil (FLOT) in Patients With Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Pilot Study of Perioperative Docetaxel, Oxaliplatin, and 5-Fluorouracil (FLOT) in Gastroesophageal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dr. Thierry Alcindor, MD, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGH-TA-01 / McG 1319
Record Dates: First submitted 2013-08-23; First posted 2013-08-30 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Gastric Adenocarcinoma; Esophageal Adenocarcinoma
Keywords: gastric; esophageal; adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Adenocarcinoma | interventions — Fluorouracil; Oxaliplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLOT chemotherapy (Other): Chemotherapy to be administered every 2 weeks for 4 cycles, before surgery. Then 4 more cycles will be given after surgery, at 2-week intervals.
  5-FU 2600 mg IV/m2 in continuous infusion Leucovorin 200 mg IV/m2 Oxaliplatin 85 mg IV/m2 Docetaxel 50 mg IV/m2
  Interventions: Drug: FLOT (5-fluorouracil, oxaliplatin, docetaxel)

INTERVENTIONS:
Drug: FLOT (5-fluorouracil, oxaliplatin, docetaxel) — Administration of FLOT chemotherapy before and after surgery
  Other Names: Oxaliplatin: Eloxatin; Docetaxel: Taxotere

SUMMARY:
Gastric or gastroesophageal junction adenocarcinoma is commonly treated with chemotherapy before and after surgery. The chemotherapy regimen used in our institution, called DCF (docetaxel,cisplatic, 5-fluorouracil) is active, resulting in tumor reduction and dysphagia relief. however, it is toxic, causing approximately half of patients severe inflammation of the mucosa (lining) of the mouth and gut. This results, in turn, in mouth sores, vomiting and diarrhea. Similar regimen called FLOT (5-FU, oxaliplatin,docetaxel) appears to be at least equally active, but less toxic.

Our ultimate plan is to perform a randomized comparison of DCF and FLOT. Before embarking upon this, we are conducting this pilot trial in 10 subjects with the FLOT regimen. If less than 5 patients develop severe mouth sores, vomiting or diarrhea, plans will be made to proceed with the next trial, a randomized comparison of DCF and FLOT

DETAILED DESCRIPTION:
Data about occurrence of diarrhea and mouth sores will be recorded through the use of quality-of-life questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of adenocarcinoma of the stomach, gastro-esophageal junction (GEJ), or lower third of the esophagus.
* The tumor must be deemed by the team to be potentially resectable. This includes imaging studies (detailed below) to clinically stage the tumor and rule out the presence of metastatic disease, and includes a preoperative laparoscopic evaluation.
* Stage IB (T1N1 only), II, IIIA, IIIB, and IV (T4N1 only)
* Life expectancy greater than 3 months
* ECOG performance status of 0-2 (i.e. restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work).
* Adequate hematologic reserve: Platelet count greater than or equal to 100,000 microlitre, WBC greater than or equal to 2000 microlitre,
* Creatinine clearance greater than or equal to 30 ml/min, AST & ALT less than or equal to 2 ULN, Alkaline phosphatase less than or equal to 2.5 ULN, bilirubin less than or equal ULN

Exclusion Criteria:

* Prior systemic therapy for gastric cancer
* Prior docetaxel-containing chemotherapy
* Pre-existing medical conditions precluding treatment, including any contraindication for major surgery
* Pregnancy or lactating mothers. Women of childbearing age must use contraception during and for 3 months following treatment
* Inability to give informed consent
* Inability to maintain nutrition by oral consumption of food alone must have additional enteral feeding.
* Macroscopic disease noted at laparoscopy
* ECOG peformance status of 3 or higher
* Unwillingness to undergo investigations and/or treatment as outlined on the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Rate of severe gastrointestinal toxicity (grade 3-4) stomatitis or diarrhea) in the preoperative setting. | One year
  Measurement through quality-of-life questionnaire

SECONDARY OUTCOMES:
Improvement of dysphagia score | 1 and 2 months
  Measurement through dysphagia score

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Alcindor, MD, MSc, Study Chair — McGill University
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada